CLINICAL TRIAL: NCT03249974
Title: A Comparative Study on the Accuracy, Ease of Use and Skin Reactions Between the Enlite Sensor With Guardian 2 Link Transmitter and the FreeStyle Libre Flash Glucose Sensor
Brief Title: Comparison Between Enlite and Flash Glucose Monitoring
Status: Completed | Type: Observational
Sponsor: Jessa Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: JessaH_B243201732756
Record Dates: First submitted 2017-07-10; First posted 2017-08-15 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2017-07

CONDITIONS: Type1 Diabetes Mellitus
Keywords: Enlite glucose monitoring; accuracy; usability; skin reactions; type 1 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Target group: Children (5 to 18 years) with type 1 diabetes mellitus treated with an insulin pump and wearing a FreeStyle Flash Libre glucosesensor will switch to the Enlite sensor communicating with Minimed 640G pump
  Interventions: Device: Enlite sensor communicating with Minimed 640G pump

INTERVENTIONS:
Device: Enlite sensor communicating with Minimed 640G pump — Children (5 to 18 years) with type 1 diabetes mellitus treated with an insulin pump and wearing a FreeStyle Flash Libre glucosesensor will switch to the Enlite sensor communicating with Minimed 640G pump

SUMMARY:
1. The accuracy of the sensors (Flash vs Enlite glucose monitoring) will be evaluated with a standardized breakfast test. Patients receive a standardized breakfast. The usual insulin bolus will be administered at breakfast. After breakfast, a venous blood sample is taken for 2 hours every 15 minutes to determine the blood sugar. At the same time, the glucose value shown by the sensors will be noted. A comparison of the blood glucose value with the data recorded by the sensor can evaluate the accuracy of the sensor and also estimate the lag-time between the sensor glucose and the venous glucose.
2. Patient satisfaction will be evaluated using a questionnaire that will be completed after the Enlite sensor has been worn for 1 month.
3. The development of skin reactions will be checked by a short questionnaire, supplemented with a picture of possible skin phenomena.
4. The data recorded by the FreeStyle sensor (average glucose,% above target,% within target,% under target, amount of hypoglycemia) in the month prior to sensor switching will be compared to the same data recorded by the Enlite sensor during the first month of use.

ELIGIBILITY:
Inclusion Criteria:

* Children (5 to 18 years)
* Diagnosis of type 1 diabetes mellitus
* Treatment is an insulin pump and wearing a FreeStyle Flash Libre glucosesensor

Exclusion Criteria:

-

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children (5 to 18 years) with type 1 diabetes mellitus treated with an insulin pump and wearing a FreeStyle Flash Libre glucosesensor
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-07-04 (Actual)

PRIMARY OUTCOMES:
Accuracy of Enlite sensor | 2 hours
  The accuracy of the sensors (flash vs enlite glucose monitoring) will be evaluated with a standardized breakfast test. Patients receive a standardized breakfast. The usual insulin bolus will be administered at breakfast. After breakfast, a venous blood sample is taken for 2 hours every 15 minutes to determine the blood sugar. At the same time, the glucose value shown by the sensors will be noted. A comparison of the blood glucose value with the data recorded by the sensor can evaluate the accuracy of the sensor and also estimate the lag-time between the sensor glucose and the venous glucose.

SECONDARY OUTCOMES:
Usability of Enlite sensor | 1 month
  Patient satisfaction will be evaluated using a questionnaire that will be completed after the Enlite sensor has been worn for 1 month.
skin reactions wih Enlite sensor | 1 month
  The development of skin reactions will be checked by a short questionnaire, supplemented with a picture of possible skin phenomena.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Massa, MD, PhD, Principal Investigator — Jessa Hospital, hasselt, Belgium
Locations (1):
- Jessa Hospital, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: No